CLINICAL TRIAL: NCT04881214
Title: Impact of COVID-19 Pneumonia on Pulmonary Physiology, Health-related Quality of Life and Benefit of a Rehabilitation Program (COVISQAR)
Brief Title: COVID-19 Pneumonia: Pulmonary Physiology, Health-related Quality of Life and Benefit of a Rehabilitation Program
Acronym: COVISQAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Principal Investigator, Frédéric Lador, MD-PhD, Medical doctor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001457
Record Dates: First submitted 2020-07-03; First posted 2021-05-11 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Covid19 Pneumonia; Chronic Thromboembolic Pulmonary Hypertension; Myopathy; Restrictive Lung Disease
Keywords: COVID-19; cardiopulmonary rehabilitation; spirometry; thromboembolic disease; non-invasive cardiac output
MeSH Terms: conditions — Muscular Diseases; COVID-19; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in this arm will receive standard of care
- Pulmonary Rehabilitation (Experimental): Patients will undergo a 12-weeks Pulmonary rehabilitation program. It will include 3 sessions of supervised exercise per week, as initially proposed on COPD patients. Patients will exercise on electromagnetically braked cycle ergometers for 45 min by alternating 30-s exercise intervals at 100% of peak-work rate estimated during the initial incremental test, with 30-s rest periods. Total workload will be increased (by 5%) on a weekly basis. Strength training of lower and upper limbs, will also be included.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — pulmonary rehabilitation for 12 weeks, 3 times a week. control will take place at 3, 6 and 12 months
  Arms: Pulmonary Rehabilitation

SUMMARY:
The pathophysiological processes involved in COVID-19 pneumonia are not fully understood. Specific alterations of the airways, lung parenchyma and pulmonary vascular tree could explain a severe ventilation/perfusion heterogeneity resulting in severe hypoxemia during the active phase of the disease. Additional skeletal muscle impairment related to systemic inflammation may also explain persisting symptoms in the follow-up phase. The first aim of the present project is to explore these different processes by evaluating the impact of the COVID-19 pneumonia on exercise capacity, pulmonary function and perfusion by a physiological and radiologic study. An ambulatory pulmonary rehabilitation will also be studied to assess its impact on the physiological parameter mentioned and the health-related quality of life questionnaire as a potential long-term treatment. The investigators propose a single center randomized controlled study at the University Hospitals of Geneva. 60 adult patients having suffered a hypoxemic COVID-19 pneumonia with persistent symptoms at 3-months after hospital discharge will be included. A functional and physiological study will be performed, including a six-minute walk test, pulmonary function testing, diffusing capacity for carbon monoxide, maximal inspiratory pressure and sniff nasal inspiratory pressure. Those with at least one abnormal value will be invited to fill the Saint Georges Respiratory Questionnaire, the Short Form 36 and the Hospital Anxiety and Depression Scale and will undergo a chest dual energy computed tomography (DECT), a cardiopulmonary exercise testing with non-invasive cardiac output and stroke volume evaluation and an evaluation of the pulmonary shunt by hyperoxia (100% oxygen breathing) at rest and during light effort. Then patients will be randomized on a 1:1 basis for pulmonary rehabilitation program or usual care. All work-up except DECT will be repeated at 6 and 12 months after hospital discharge. The investigators hypothesize that our study will allow a better understanding of pathophysiological mechanisms involved in COVID-19. This will potentially determine therapeutic target for patients with persisting symptoms and functional decay after COVID-19. The investigators also expect to see an improvement of exercise capacity and physiological parameters in the pulmonary rehabilitation group, as compared to the control group, suggesting pulmonary rehabilitation as a possible long-term treatment of this condition.

DETAILED DESCRIPTION:
COVID-19 is an emerging pandemic disease caused by a novel coronavirus (SARS-CoV-2) since December 2019. This condition may be associated with a severe pneumonia and an acute respiratory distress syndrome (ARDS) resulting in a high mortality and morbidity.A standardized follow up of COVID-19 patients after discharge from Geneva University Hospitals (Covicare) was implemented since March 29th 2020 by the divisions of infectious disease and respiratory medicine, in association with the primary care medicine department. A follow-up is ensured until one month after discharge. All patients are registered in a database (REDCapTM,Tennessee, USA).

The pathophysiological mechanisms of ARDS in COVID-19 and its long-term consequences on respiratory and cardiovascular systems remain unclear. Several histopathological studies have demonstrated occurrence of interstitial lung disease. Furthermore, there are some reports of associated endothelitis, thrombosis in the microcirculation5 and a high prevalence of venous thrombo-embolic events in ICU admitted patients, with pulmonary embolism accounting for 85% of those events.Both these changes contribute to increase heterogeneity of ventilation - perfusion ratio (VA/Q), thereby widening the alveolar - arterial oxygen gradient, and thus causing serious hypoxaemia, with remarkable fall of arterial oxygen saturation (SaO2). Finally, the interstitial pneumopathy may cause a persisting reduction of lung diffusing capacity for carbon monoxide (DLCO), further decreasing SaO2 even after recovery from COVID-19 pneumonia.

Chest Dual-Energy Computed Tomography (DECT) enables a combined functional and morphological analysis of the lung in a single and simple acquisition. Because of the attenuation properties of iodine at two different photon energies (80 and 140kV), DECT is able to reveal pulmonary blood volume distribution and generate color-coded pulmonary iodine volume maps, corresponding to the pulmonary perfusion. These pulmonary perfusion maps allow a qualitative analysis of the perfusion.Furthermore, the iodine concentration of the lung confers an objective and quantitative regional analysis of the perfusion. In comparison with a conventional CT, no additional intravenous iodine contrast medium injection or radiation doses are needed; a functional image processing is simply added. We recently demonstrated how DECT may help to define lung perfusion changes after therapeutic measures in patients with chronic obstructive pulmonary disease. Moreover, DECT offers an excellent correlation with perfusion scintigraphy (V/Q scan). DECT also offers a superior anatomic and functional comprehension by simultaneously recording the vascular anatomy, parenchymal morphology, and functional perfusion. Consequently, DECT may provide important information both on persisting parenchymal and perfusion alteration after COVID-19.

In addition to the pulmonary component, the systemic inflammation state due to the concurring "cytokine storm syndrome" may have an important role in the development of neuromuscular alterations, independently of direct consequences of hospitalization in intensive care unit. Neuromuscular alterations concur with lung function impairment in compromising the functional state of the patient. As a consequence, we ought to expect a reduction of physical exercise capacity, which is normally determined by a VO2max measurement during cardiopulmonary exercise test (CPET) and by means of the six-minute walk test (6MWT).

Moreover, it is well described that ARDS is associated with a significant long-term morbidity. At one year, 80% of ARDS survivors have a reduced diffusing capacity and 20% suffer from an airflow obstruction. 35% of patients have an exercise limitation based on the 6MWT at two years. Moreover, impairment in lung function, musculoskeletal dysfunction and functional limitation are linked to health-related quality of life (HRQL) decrement.

Studies from a cohort of patients who suffered from ARDS due to SARS-CoV-1 in 2002 showed a positive correlation between lung function and the HRQL physical functioning domain. Distance performed during 6MWT correlated also with almost all Short Form Health Survey-36 (SF-36) domains. Furthermore, mood disorders are commonly described in ARDS survivors, with studies reporting up to 50% of depression at one year in this population. Depression and anxiety are themselves associated with lower HRQL scores.

Pulmonary rehabilitation has been shown to improve HRQL, maximal exercise capacity and 6MWD in chronic pulmonary disease. It was also shown that 2 months of ambulatory pulmonary rehabilitation improved pulmonary function and the St. George's Respiratory Questionnaire (SGRQ) at 3 and 6 months post-discharge following recovery from ARDS due to severe influenza A (H1N1 in 2009) pneumonitis.

The purpose of this study is 1/ to explore the long-term impact of COVID-19 on physiological respiratory parameters, functional capacity, HRQL and mood disturbances ; 2/ to assess the benefit of a pulmonary rehabilitation program on these outcomes through a randomized-control study, and 3/ to determine the contribution of DECT to the understanding of the pathophysiological alterations in patients with functional sequelae of COVID-19 infection.

ELIGIBILITY:
Patients will be eligible for inclusion if they fulfil all the following criteria:

* Patients aged ≥ 18 years.
* Confirmed diagnosis of SARS-Cov-2 infection by nasal swab, other viral sample (i.e. sputum, bronchoalveolar lavage) or Chest imaging suggestive of SARS-CoV-2 pneumonia (Chest X-ray or CT-scan).
* Requirement for oxygen supplementation.
* Persistent respiratory symptoms (i.e. dyspnoea, cough) or asthenia.
* Abnormal 6MWT at 3 months (distance < 90% predicted or desaturation ≥ 3% or Borg >5) and/or abnormal lung function as described by the international recommendations

Patients will be excluded if they:

* Already had existing severe and symptomatic pulmonary condition before COVID-19 pneumonia
* Are unable to execute the different tests and surveys because of cognitive or physical limitations.
* Are already included in a structured rehabilitation program
* Have comorbidities with a life expectancy of less than 12 months.
* Any relevant acute medical disorder/acute disease state judged by the investigators as likely to represent a risk for the patient to fulfil a rehabilitation program or requiring urgent investigations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of ambulatory pulmonary rehabilitation in health related quality of life | 12 months
  St George's Respiratory questionnaire change (units). Scores range from 0 to 100, with higher scores indicating more limitations

SECONDARY OUTCOMES:
Long-term consequences of COVID-19 pneumonia on VEMS | 12 months
  Change in VEMS (L, % predicted)
Long-term consequences of COVID-19 pneumonia on Vital Capacity | 12 months
  Change in Vital Capacity (L, % predicted)
Long-term consequences of COVID-19 pneumonia on Total Lung Capacity | 12 months
  Change in Total Lung Capacity (L, % predicted)
Long-term consequences of COVID-19 pneumonia on diffusion capacity of CO | 12 months
  Change in diffusion capacity of CO (ml/min/kPa, % predicted)
long-term consequences of COVID-19 pneumonia on Vital Capacity (VC) | 12 months
  absolute value (liters) measured at inclusion and at the end of the study period with spirometry
long-term consequences of COVID-19 pneumonia on total lung capacity (TLC) | 12 months
  absolute value (liters) measured at inclusion and at the end of the study period with plethysmography
long-term consequences of COVID-19 pneumonia on diffusing capacity for carbon monoxide (DLCO) | 12 months
  absolute value (ml/min/kPa) measured at inclusion and at the end of the study period with plethysmography
Incidence of interstitial lung disease and/or images suggestive of abnormalities in the pulmonary circulation. | 3 months
  Evaluated with a chest dual energy Computed Tomography: presence of honeycombing, bronchiectasis or acute or chronic thromboembolism.
Effect of COVID-19 pneumonia on The Short Form 36 (SF-36) questionnaire score | 12 months
  measured at inclusion and at the end of the study. Score from 0 (poor health) to 100 (perfect health)
Effect of COVID-19 pneumonia on Hospital Anxiety and Depression Scale (HADS) score | 12 months
  measured at inclusion and at the end of the study. . Each of them is coded From 0 to 3, with a score varying from 0 to 21
Effect of pulmonary rehabilitation in VO2 max during cardiopulmonary exercise testing (CPET) | 3,6 and 12 months
  Change in VO2 max (ml/min/kg)
Effect of pulmonary rehabilitation in power during cardiopulmonary exercise testing (CPET) | 3,6 and 12 months
  Change in power max (Watts)
Effect of pulmonary rehabilitation in ventilation during cardiopulmonary exercise testing (CPET) | 3,6 and 12 months
  Change in ventilation (L/min)
Effect of pulmonary rehabilitation in Tidal Volume during cardiopulmonary exercise testing (CPET) | 3,6 and 12 months
  Change in Tidal Volume (L)
Effect of pulmonary rehabilitation in 6 minutes walk test distance | 3,6 and 12 months
  Change in meters
Effect of pulmonary rehabilitation in 6 minutes walk test dyspnea | 3,6 and 12 months
  Change in self reported Borg dyspnea
Effect of pulmonary rehabilitation in cardiac output during CPET | 3,6 and 12 months
  ANOVA comparison of cardiac output with 2 non-invasive measurement of cardiac output
Evaluation of COVID-19 impact in pulmonary shunt effect | 2,6 and 12 months
  Change in pulmonary shunt (delta kPa)

CONTACTS AND LOCATIONS:
Overall Officials: Lador Frédéric, MD-PHD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finegan O, Fonseca S, Guyomarc'h P, Morcillo Mendez MD, Rodriguez Gonzalez J, Tidball-Binz M, Winter KA; ICRC Advisory Group on the Management of COVID-19 Related Fatalities. International Committee of the Red Cross (ICRC): General guidance for the management of the dead related to COVID-19. Forensic Sci Int Synerg. 2020 Mar 31;2:129-137. doi: 10.1016/j.fsisyn.2020.03.007. eCollection 2020. PMID 32412013
- [Background] Correction to Lancet Respir Med 2020; 8: 420-22. Lancet Respir Med. 2020 Apr;8(4):e26. doi: 10.1016/S2213-2600(20)30085-0. Epub 2020 Feb 25. No abstract available. PMID 32109426
- [Background] Tian S, Hu W, Niu L, Liu H, Xu H, Xiao SY. Pulmonary Pathology of Early-Phase 2019 Novel Coronavirus (COVID-19) Pneumonia in Two Patients With Lung Cancer. J Thorac Oncol. 2020 May;15(5):700-704. doi: 10.1016/j.jtho.2020.02.010. Epub 2020 Feb 28. PMID 32114094
- [Background] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Derived] Guerreiro I, Bringard A, Nehme M, Guessous I, Benzakour L, Juillet De Saint Lager-Lucas A, Taboni A, Lador F. Exercise ventilatory response after COVID-19: comparison between ambulatory and hospitalized patients. Am J Physiol Lung Cell Mol Physiol. 2023 Dec 1;325(6):L756-L764. doi: 10.1152/ajplung.00142.2023. Epub 2023 Oct 24. PMID 37874657